CLINICAL TRIAL: NCT00409422
Title: Effects of a Comprehensive Weight Management Program on Obese Adolescents and Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sonia Caprio, MD, Yale University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIC 15994
Record Dates: First submitted 2006-12-06; First posted 2006-12-08 (Estimated); Last update posted 2008-06-24 (Estimated); Status verified 2008-06

CONDITIONS: Pediatric Obesity; Insulin Resistance; Hyperinsulinemia
Keywords: pediatric obesity; overweight; insulin resistance; hyperinsulinemia; weight management program; family-based
MeSH Terms: conditions — Pediatric Obesity; Insulin Resistance; Hyperinsulinism; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: weight management program

SUMMARY:
To compare anthropometric and metabolic effects of a comprehensive weight management program on obese adolescents and children in comparison to regular clinical weight management visits.

DETAILED DESCRIPTION:
Patients are randomized (2:1) to either the intensive or standard treatment (control). Those who get randomized into the intensive group go to a family-based weight management program, including exercise, nutrition, behavior modification, and parenting classes. The intensive group is further randomized into a diet or non-dieting class to compare the outcomes of two different nutrition intervention methods. These classes meet twice per week (exercise twice per week and nutrition/behavior modification once per week)for first six months and then only twice per month during last six months. An exercise physiologist supervises the exercise component, which involves 45 minutes of aerobic activity (targeted at 65 to 80 percent of the subject's estimated maximum heart rate. A registered dietitian facilitates the nutrition and behavior component. A social worker facilitates parent classes when the children have a behavior modification topic in their class (parents only attend nutrition sessions). Those who get randomized into the control group go to clinic visits every 6 months. Intervention subjects go to clinic, as well, every 6 months to obtain the same measurements as the controls (weight, BMI, % fat, fasting insulin, fasting glucose, lipids, blood pressure).

ELIGIBILITY:
Inclusion Criteria:

* Ages 8-16 years old
* BMI >95th percentile for age/gender based on CDC
* Both primary caregiver/parent and child must agree to participate in the nutrition classes

Exclusion Criteria:

* endocrinopathies, including hypothyroidism and diabetes
* Psychiatric disorders that will interfere with ability to complete follow-up and adherence to protocol
* Any behavioral or psychosocial issue that will interfere with subject's completion of program, including eating disorder.
* Any use of medication (steroids, for ex.) that contributes to excess adiposity.
* Any use of pharmacological intervention for weight management, including prescription medications, over-the-counter medications, or herbal supplements.
* Any concurrent membership in a weight management program.
* Inability or unwillingness of parent to accompany the child to nutrition classes.
* Pregnancy

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200
Dates: Start 2002-05; Primary Completion 2006-10 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
weight | 6 months and 1 year
body mass index | 6 months and 1 year
% body fat | 6 months and 1 year
lipids | 6 months and 1 year
blood pressure | 6 months and 1 year
glucose | 6 months and 1 year
insulin | 6 months and 1 year
HOMA index | 6 months and 1 year

SECONDARY OUTCOMES:
planned to compare dieting with non-dieting approach in weight management group | 6 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Caprio, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Savoye M, Shaw M, Dziura J, Tamborlane WV, Rose P, Guandalini C, Goldberg-Gell R, Burgert TS, Cali AM, Weiss R, Caprio S. Effects of a weight management program on body composition and metabolic parameters in overweight children: a randomized controlled trial. JAMA. 2007 Jun 27;297(24):2697-704. doi: 10.1001/jama.297.24.2697. PMID 17595270